CLINICAL TRIAL: NCT00090974
Title: Quality Of Life Companion Study For JMA27 (NCIC-MA.27): A Randomized Phase III Trial Of Exemestane Versus Anastrozole With Or Without Celecoxib In Postmenopausal Women With Receptor Positive Primary Breast Cancer
Brief Title: Quality of Life in Postmenopausal Women Who Are Receiving Either Exemestane or Anastrozole With or Without Celecoxib for Stage I, Stage II, or Stage IIIA Primary Breast Cancer
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Other Study IDs: CDR0000380937; U10CA021115 (NIH); ECOG-E1Z03; CAN-NCIC-E1Z03
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Quality-of-life assessment in postmenopausal women who are receiving hormone therapy for breast cancer may help to determine the effects of treatment on these patients and may improve the quality of life for future breast cancer patients.

PURPOSE: This clinical trial is studying quality of life of postmenopausal women who are receiving either exemestane or anastrozole with or without celecoxib for stage I, stage II, or stage IIIA primary breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare treatment-related symptoms using the Functional Assessment of Cancer Therapy-Endocrine Symptoms (FACT-ES) questionnaire in postmenopausal women with receptor-positive stage I, II, or IIIA primary breast cancer undergoing treatment with exemestane vs anastrozole with or without celecoxib on protocol CAN-NCIC-MA27.

Secondary

* Compare health-related quality of life using the FACT-ES questionnaire in patients treated with these regimens.
* Determine the extent to which differences in treatment-emergent symptoms affect overall quality of life in patients treated with these regimens.

OUTLINE: This is a multicenter, companion study. Patients receive treatment on CAN-NCIC-MA27.

Health-related quality of life and treatment-related symptoms are assessed using the Functional Assessment of Cancer Therapy-Endocrine Symptoms (FACT-ES) questionnaire at baseline and at 3, 6, 12, and 24 months.

PROJECTED ACCRUAL: A total of 1,253 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * pT1-3; pNX, pN0-2 or pN3*; M0 NOTE: *Only when the sole basis for this classification is the presence of 10 or more involved axillary lymph nodes
* Registered on protocol CAN-NCIC-MA27 within the past week
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive by immunohistochemistry or tumor receptor content ≥ 10 fmol/mg protein
  * At least 1 tumor must be receptor-positive in patients with bilateral breast cancer

PATIENT CHARACTERISTICS:

Age

* Postmenopausal

Performance status

* ECOG 0-2

Sex

* Female

Menopausal status

* Postmenopausal

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Able to read, understand, and complete quality of life questionnaires

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 0 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-01-26 (Actual); Primary Completion 2013-01-30 (Actual); Study Completion 2013-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Wagner, MD, Study Chair — Robert H. Lurie Cancer Center; Paul E. Goss, MD, PhD, Study Chair — Massachusetts General Hospital
Locations (224):
- United States (224):
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Banner Thunderbird Medical Center, Phoenix, Arizona
  - North Bay Cancer Center, Fairfield, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Memorial Medical Center Cancer Services, Modesto, California
  - Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - John B. Amos Community Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Delnor Community Hospital - Geneva, Geneva, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology-Oncology Associates at June E. Nylen Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, P.A. - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, P.A. - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, P.A. - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, P.A. - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - Cancer Center of Kansas, P.A. - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, P.A. - Salina, Salina, Kansas
  - Cancer Center of Kansas, P.A. - Wellington, Wellington, Kansas
  - Associates in Womens Health, P.A. - North Review, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Winfield, Winfield, Kansas
  - Lawrence Memorial Hospital of Medford, Medford, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, P.C., Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Oncology Care Associates, P.L.L.C., Saint Joseph, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Cancer Care Center at St. Luke's Hospital, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine Associates of Bozeman, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Community Oncology Group - Independence, Independence, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center Oncology Unit, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Toledo Surgical Specialists, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Valley Medical Center, Renton, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Solomon SD, Wittes J, Finn PV, Fowler R, Viner J, Bertagnolli MM, Arber N, Levin B, Meinert CL, Martin B, Pater JL, Goss PE, Lance P, Obara S, Chew EY, Kim J, Arndt G, Hawk E; Cross Trial Safety Assessment Group. Cardiovascular risk of celecoxib in 6 randomized placebo-controlled trials: the cross trial safety analysis. Circulation. 2008 Apr 22;117(16):2104-13. doi: 10.1161/CIRCULATIONAHA.108.764530. Epub 2008 Mar 31. PMID 18378608